CLINICAL TRIAL: NCT02682459
Title: A Pilot, Prospective, Randomized, Open-label, Blinded Endpoint (Probe) Histopathology Trial to Assess the Effects of ACE- Inhibition Therapy on Glomerular Proliferative Lesions in Patients With Extracapillary Glomerulonephritis
Brief Title: ACE-inhibitors in Extracapillary Glomerulonephritis
Acronym: EXTRA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Monia Lorini (Other)
Collaborators: Istituto Di Ricerche Farmacologiche Mario Negri (Other)
Responsible Party: Sponsor-Investigator, Monia Lorini, EC Secretary, A.O. Ospedale Papa Giovanni XXIII
Organization: A.O. Ospedale Papa Giovanni XXIII (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EXTRA; 2015-003884-12 (EudraCT Number)
Record Dates: First submitted 2016-02-10; First posted 2016-02-15 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Extracapillary Glomerulonephritis
Keywords: Extracapillary glomerulonephritis; crescentic glomerulonephritis; rapidly progressive renal failure; chronic kidney disease; ACE-inhibitors; fibrosis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Fibrosis | interventions — Lisinopril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lisinopril (Experimental): Patients will receive, in addition to standard immunosuppressive therapy, lisinopril starting with 5 mg/day, then progressively up-titrated to reach the maximum tolerable dose (target dose) for 18 months.
  Interventions: Drug: Lisinopril
- No intervention (No Intervention): Patients will receive only the standard immunosuppressive therapy.

INTERVENTIONS:
Drug: Lisinopril
  Arms: Lisinopril

SUMMARY:
The natural course of extracapillary glomerulonephritis is severe leading to End-Stage Renal Disease (ESRD) or death in most cases. Despite immunosuppressive treatment, long-term renal outcome remains poor since active crescents usually progress to fibrotic scars with glomerular occlusion and disruption.In experimental models Angiotensin Converting Enzyme (ACE)-inhibitor therapy targeting the over-expression of angiotensin type 1 (AT1) receptors, that are responsible for dysregulated proliferation of parietal cell progenitors, blocks the formation of crescents and their fibrotic evolution. Should these drugs have similar effects in humans, ACE-inhibitor therapy on top of standard immunosuppression might be instrumental to prevent ESRD and promote renal function recovery in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Rapidly progressive renal failure associated with acute nephritic syndrome and/or nephrotic syndrome;
* Histology evidence of extracapillary proliferation with less than 50% of sclerotic glomeruli and associated with:

  1. Type I: Anti-Glomerular Basement Membrane (GBM) antibody glomerulonephritis,
  2. Type II: Pauci-immune vasculitis or Anti Neutrophil Cytoplasmic Antibody (ANCA) associated vasculitis;
  3. Type III: Immune-complex mediated glomerular diseases: Proliferative lupus nephritis (LN), IgA nephropathy (IgAN)/ Schönlein-Henoch purpura, Type I membranoproliferative glomerulonephropathy (MPGN), Primary or secondary membranous nephropathy (MN), Primary or idiopathic immune complex glomerulonephritis.
* Clinical indication to immunosuppressive therapy;
* No specific indication to treatment with Renin Angiotensin System (RAS) inhibitors such as heart failure or coronary ischemic disease;
* Written informed consent.

Exclusion Criteria:

* Pre-existing advanced chronic renal failure (creatinine clearance less than 20 ml/min/1.73m2);
* Evidence of B or C virus active infection;
* HIV infection;
* Recent diagnosis of malignancy;
* Prolonged bleeding time and any other contraindication to kidney biopsy evaluation;
* Any specific contraindication to ACE inhibitor therapy (that is: history of angioedema or other treatment-related serious adverse events);
* Pregnancy or lactating;
* Women of childbearing potential without following a scientifically accepted form of contraception;
* Inability to understand the risks and benefit of the study or evidence of an uncooperative attitude;
* Legal incapacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2016-02; Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The extent of extracapillary proliferation on light microscopy, measured as % of total glomeruli with proliferative lesions at post-treatment repeat biopsy. | Changes from baseline and 6 and 18 month.

SECONDARY OUTCOMES:
Expression of parietal cell proliferation markers at glomerular level, graded on a scale of 0 to 3 (0: no staining, 1: mild, 2: moderate, 3: strong diffuse | Changes from baseline and 6 and 18 month.
Number of fibrosclerotic crescents | Changes from baseline and 6 and 18 month.
Glomerular Filtration Rate (GFR) measured by iohexol plasma clearance | Changes from baseline and 6, 12 and 18 month.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Centro di Ricerche Cliniche per le Malattie Rare Aldo e Cele Daccò, Ranica, Bergamo
  - ASST Papa Giovanni XXIII, Bergamo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hruskova Z, Honsova E, Berden AE, Rychlik I, Lanska V, Zabka J, Bajema IM, Tesar V. Repeat protocol renal biopsy in ANCA-associated renal vasculitis. Nephrol Dial Transplant. 2014 Sep;29(9):1728-32. doi: 10.1093/ndt/gfu042. Epub 2014 Feb 26. PMID 24578468
- [Background] Smeets B, Angelotti ML, Rizzo P, Dijkman H, Lazzeri E, Mooren F, Ballerini L, Parente E, Sagrinati C, Mazzinghi B, Ronconi E, Becherucci F, Benigni A, Steenbergen E, Lasagni L, Remuzzi G, Wetzels J, Romagnani P. Renal progenitor cells contribute to hyperplastic lesions of podocytopathies and crescentic glomerulonephritis. J Am Soc Nephrol. 2009 Dec;20(12):2593-603. doi: 10.1681/ASN.2009020132. Epub 2009 Oct 29. PMID 19875807
- [Background] Benigni A, Morigi M, Rizzo P, Gagliardini E, Rota C, Abbate M, Ghezzi S, Remuzzi A, Remuzzi G. Inhibiting angiotensin-converting enzyme promotes renal repair by limiting progenitor cell proliferation and restoring the glomerular architecture. Am J Pathol. 2011 Aug;179(2):628-38. doi: 10.1016/j.ajpath.2011.04.003. Epub 2011 Jun 2. PMID 21718676